CLINICAL TRIAL: NCT02957175
Title: Immunophenotyping of Patients Undergoing Open Heart Surgery to Assess Their Susceptibility of Developing a Systemic Inflammatory Response Syndrome (SIRS)
Brief Title: Immunophenotyping of Patients With Postoperative SIRS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bonn (Other)
Responsible Party: Principal Investigator, Dr. Christian Bode, Principal Investigator, University of Bonn
Other Study IDs: BOST-001
Record Dates: First submitted 2016-09-30; First posted 2016-11-07 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: Immunophenotyping; Perioperative Care; Innate Immunity; Cardiac Surgical Procedures
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome | interventions — Immunophenotyping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and Leukocytes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients that develop SIRS: Immunophenotyping of patients that develop SIRS after heart surgery
  Interventions: Other: Immunophenotyping
- Patients that develop no SIRS: Immunophenotyping of patients that develop no SIRS after heart surgery
  Interventions: Other: Immunophenotyping

INTERVENTIONS:
Other: Immunophenotyping — Multiplex assays for screening pro- and anti-inflammatory markers and RNA will be analysed using a next generation sequencing approach

SUMMARY:
The purpose of this study is to develop an immune-phenotype based prediction of postoperative SIRS in patients undergoing open heart surgery.

DETAILED DESCRIPTION:
The study will have a pre-, intra and postoperative phase in which several demographic and clinical variables will be assessed. The samples for the immunophenotypic analysis will be drawn directly after induction of anesthesia and at various time points after end of surgery. The diagnosis of SIRS will be made during routine clinical visits on the first seven postoperative days using the Sepsis-related Organ Failure Assessment score (SOFA-score). The patients will be followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Informed consent of the patient
* Patient undergoing a open heart surgery using a cardiopulmonary bypass

Exclusion Criteria:

* Age < 18 years
* Missing informed consent
* Renal failure
* Liver failure
* Neurodegenerative disease
* Malignancies
* Immune therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing open heart surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with SIRS as assessed by SOFA-Score | 30 days
  The study investigates the relationship between the intra-individual inflammatory patterns in patients with uncomplicated (no SIRS) and complicated postoperative courses (SIRS) after open heart surgery.
  The diagnosis of SIRS will be made by using the Sepsis-related Organ Failure Assessment score (SOFA-score). Patients with an increase in SOFA-score >3 are considered to have SIRS.

SECONDARY OUTCOMES:
Number of participants with need for renal replacement therapy because of acute kidney failure (AKIN classification) | 30 days
Number of participants with infection as assessed by microbiological, serological and radiological examination | 30 days
Number of participants with postoperative delir as assessed by CAM-ICU | 30 days
Number of participants with myocardial injury as assessed by troponine and CK-MB serum levels | 30 days
Number of participants with new atrial fibrillation as assessed by ECG | 30 days
Length of stay in ICU | 30 days
Length of stay in hospital | 30 days
In-hospital mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Eicke Latz, MD, PhD, Study Chair — Institute of Innate Immunity; Christian Bode, MD, Study Chair — Department of Anesthesia and Critical Care Medicine; Folkert M Steinhagen, MD, Principal Investigator — Department of Anesthesia and Critical Care Medicine
Locations (1):
- University Hospital Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.kai.uni-bonn.de/